CLINICAL TRIAL: NCT03876444
Title: Intravenous Methylprednisolone Versus High Dose Oral Prednisolone for the Treatment of Infantile Spasms: a Randomized Open-labelled Trial
Brief Title: Intravenous Methylprednisolone Versus Oral Prednisolone for Infantile Spasms
Acronym: MPIV
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suvasini Sharma (Other Government)
Responsible Party: Sponsor-Investigator, Suvasini Sharma, Associate Professor, Lady Hardinge Medical College
Organization: Lady Hardinge Medical College (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MethylpredIV
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Infantile Spasm
Keywords: Hypsarrythmia; Methylprednisolone; Prednisolone
MeSH Terms: conditions — Spasms, Infantile

STUDY DESIGN:
Intervention Model Description: Open label Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Pulse intravenous methylprednisolone (30 mg / kg for 3 days) followed by 1-week taper of oral prednisolone Day 1-3 Intravenous Methylprednisolone in dose of 30 mg/kg/day Day 4-6 Oral Prednisolone in dose of 2mg/kg/day Day 7-10 Oral Prednisolone in dose of 1mg/kg/day
  Interventions: Drug: Intravenous Methylprednisolone
- Control (Active Comparator): Oral prednisolone (4 mg/kg/day) for 2 weeks followed by tapering over 2 weeks Day 1-14 (2 weeks): dose 4mg/kg/day Day 15-21 (1 weeks): 2mg/kg/day Day 22-28 (1 weeks): 1mg/kg/day
  Interventions: Drug: Oral Pednisolone

INTERVENTIONS:
Drug: Intravenous Methylprednisolone — Intravenous Methylprednisolone will be used in the intervention group
  Arms: Intervention arm
Drug: Oral Pednisolone — Oral Prednisolone will be used in the Control Group
  Arms: Control

SUMMARY:
Infantile Spasms (IS) are classically refractory to the usual antiepileptic drugs and often pose a therapeutic challenge. Since, there is associated significant morbidity, much effort has been directed over the past years to evaluate the role of various anticonvulsants in the management of IS. High dose oral prednisolone has been shown to cause early cessation of spasms and resolution of hypsarrythmia on Electroencephalogram. Recently, role of intravenous methylprednislone pulse therapy has been explored as one of the therapeutic modality in IS, in order to avoid the development of side-effects associated with prolonged oral steroid therapy and maintain long-term efficacy.However, there are no studies comparing iv methylprednisolone pulse therapy with high dose oral prednisolone..

DETAILED DESCRIPTION:
Multiple studies have subsequently used higher dose of prednisolone in infantile spasms at the weight based dosing of 4-8 mg/kg/day with a maximum dose of 60mg/day. The results have shown high rates of clinical and elecroencephalographic remission with lower relapse rates.However, a major concern related to corticosteroids, especially in infants and children, is the possible development of side effects. The most frequent ones are excessive weight gain, hyperphagia, water retention with edema, cushingoid appearance, hypertension, behavioral disturbances, increased infection susceptibility, leukopenia, electrolyte disturbances, hyperglycemia, glycosuria, impaired glucose tolerance, frank diabetes and sleep disorders. Furthermore, long-term side effects such as hypothalamus-pituitary axis suppression, psychosis, osteoporosis, nephrocalcinosis, brain atrophy, cataracts and, in children, growth retardation, have also been reported.

Recently, role of intravenous methylprednislone pulse therapy has been explored as one of the therapeutic modality in IS, in order to avoid the development of side-effects associated with prolonged oral steroid therapy and maintain long-term efficacy. There have been few studies on use of iv pulse methylprednisolone in IS with small sample size, showing to a rapid improvement in EEG & cessation of spasm in majority of the infants without significant adverse effects.

Emerging evidence suggests that intravenous pulse methylprednisolone might have superior efficacy and better safety profile when compared to high dose oral prednisolone in treatment of IS.

Hence, present study aims at comparing intravenous pulse methylprednisolone versus oral prednisolone in an open label, RCT for treatment of children with IS.

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed patients aged 4 - 30 months with epileptic spasms in clusters with electroencephalographic evidence of hypsarrhythmia or its variants with or without developmental delay -

Exclusion Criteria:

1. Children with recognized progressive neurological illness will be excluded.
2. Children with chronic renal, pulmonary, cardiac or hepatic dysfunction
3. Severe malnutrition (weight for length and height for less than 3 SD for mean as per WHO growth charts)

   -

Ages: 4 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of children who achieved spasm freedom as per parental reports in both the groups | 6 weeks
  The proportion of children who achieve spasm freedom defined as no witnessed spasms on and between day 14 and day 42 as per parental reports will be evaluated in the both the groups

SECONDARY OUTCOMES:
Number of days after initiation of trial treatment on which spasms were not seen and after which response was maintained until 6 weeks (day 42) of treatment in both the groups | 6 weeks
  Number of days after initiation of trial treatment on which spasms were not seen and after which response was maintained until 6 weeks (day 42) of treatment in both the groups
Proportion of children who achieve resolution of hypsarrhythmia on electro encephalogram at 2 weeks (in all cases) and at 6 weeks (for cases with sustained clinical response) in both the groups. | 6 weeks
  Proportion of children who achieve resolution of hypsarrhythmia on electro encephalogram at 2 weeks (in all cases) and at 6 weeks (for cases with sustained clinical response) in both the groups.
Description and proportion of the adverse effects of methylprednisolone in the experimental group | 6 weeks
  Description and proportion of the adverse effects of methylprednisolone in the experimental group

CONTACTS AND LOCATIONS:
Overall Officials: Dipti Kapoor, MD, Principal Investigator — Lady Hardinge Medical College
Locations (1):
- Lady Hardinge Medical College, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kapoor D, Sharma S, Garg D, Samaddar S, Panda I, Patra B, Mukherjee SB, Pemde HK. Intravenous Methylprednisolone Versus Oral Prednisolone for West Syndrome: A Randomized Open-Label Trial. Indian J Pediatr. 2021 Aug;88(8):778-784. doi: 10.1007/s12098-020-03630-3. Epub 2021 Feb 11. PMID 33575989